CLINICAL TRIAL: NCT07241117
Title: CHEST: A Collaboration With Community HEalth Centers to Implement SmarT for Asthma
Acronym: CHEST
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Doris Duke Charitable Foundation (Other); Affinia Healthcare (Unknown); Family Care Health Centers (Unknown)
Responsible Party: Principal Investigator, James Krings, Assistant Professor of Medicine, Washington University School of Medicine
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 202507167; 5K23HL171940-02 (NIH)
Record Dates: First submitted 2025-11-07; First posted 2025-11-21 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Moderate to Severe Asthma
Keywords: asthma; SMART; moderate to severe asthma; CHEST; CHEST asthma study; asthma study; asthma action plan; implementation science; hybrid cluster; community health centers; MART; single maintenance and reliever therapy; maintenance and reliever therapy
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Intervention Model Description: This is a Phase 4, type 1 hybrid stepped-wedge cluster randomized trial conducted in six Federally Qualified Health Centers in St. Louis, Missouri. The unit of randomization is the clinic, with each site sequentially crossing over in a one-way fashion from control to intervention, allowing each to serve as its own control. The intervention is the SMART implementation bundle consisting of (1) clinician education with practice facilitation, (2) audit and feedback on prescribing, (3) patient-centered education aides, including a SMART-congruent asthma action plan, and (4) monthly operations committee meetings during implementation period. The trial proceeds in three phases: pre-implementation (baseline), active implementation (rollout), and post-implementation (sustainability/dissemination). The study population includes clinicians, staff, and patients ≥12 years with moderate-to-severe asthma.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Implementation (Experimental): The intervention is a SMART implementation bundle delivered at community health centers. It includes (1) clinician education with practice facilitation to support guideline-concordant prescribing and (2) regular audit and feedback on inhaler prescribing patterns (3) patient-centered education tools such as instructional videos and a SMART-congruent asthma action plan designed for low health literacy, and (4) operations committee meetings during the implementation period. Educational outreach is co-led by the PI and a certified asthma educator, with quarterly practice facilitation and feedback visits during the active implementation period. All materials are available in paper and digital formats, with continued access to patient tools beyond the intervention. Providers retain full autonomy over prescribing decisions
  Interventions: Behavioral: Implementation bundle
- Control (No Intervention): During this period, prescribing patterns and asthma outcomes will be observed without active implementation.

INTERVENTIONS:
Behavioral: Implementation bundle — The intervention is a SMART implementation bundle delivered in Federally Qualified Health Centers. Unlike drug trials, no medication is supplied; providers prescribe according to guidelines. The bundle includes three components: (1) clinician education with practice facilitation, (2) audit and feedback on prescribing, (3) patient education tools such as a SMART-aligned asthma action plan and videos tailored for low health literacy, and (4) operations committee meetings during the implementation period
  Arms: Active Implementation

SUMMARY:
Purpose: This study aims to improve asthma care by helping clinicians at community health centers prescribe a guideline-recommended treatment called SMART (Single Maintenance and Reliever Therapy).

The investigators will provide training and resources to clinicians, give feedback on prescribing patterns, and offer educational tools for patients and providers. The investigators will roll out these resources in stages across clinics. The study will measure how well the program helps clinicians prescribe SMART therapy and whether it reduces asthma exacerbations in patients.

DETAILED DESCRIPTION:
CHEST is a type 1 hybrid stepped-wedge cluster randomized trial wherein six federally qualified community health center clinics are randomly and iteratively selected to move in a 1-way crossover from the control group to the SMART implementation group. The primary intervention is an SMART implementation bundle, which contains three components: (1) clinician-level education on SMART with ongoing practice facilitation/supervision, (2) serial clinic- and clinician-level audit and feedback on inhaler prescribing patterns, (3) provision of a paper and online clinician- and patient-centered education aide with a SMART congruent asthma action plan designed for low health literacy patients, and (4) operations committee meetings during the implementation period

The study is conceptually split into three phases: (1) the pre-implementation (control) phase focused on development of implementation materials and baseline data gathering of prescription patterns, (2) the active implementation phase, and (3) post-implementation, which will focus on an assessment of sustainability and dissemination.

1. Pre-implementation phase: The pre-implementation phase (which will last from 12 to 24 months per clinic) is designed to be a baseline for the study. During this phase, no specific interventions will be introduced to the clinicians at participating clinics. This phase will allow the CHEST study team to collect clinic-level data on current asthma care prescription practices and asthma-related outcomes.
2. Active implementation phase: The second phase, which will last from 9 to 24 months per clinic, will begin with the introduction of the SMART implementation bundle to clinicians and staff at participating IHN clinics.
3. Post-implementation phase: The final phase of the study is introduced after the active implementation of the SMART implementation bundle is complete at all participating clinics. In the post-implementation phase, formal assessments will be conducted to evaluate the sustainment of the SMART bundle. Additionally, this phase includes efforts to disseminate the findings of the study. This encompasses analyses of the reach and impact of the dissemination efforts, as well as the practical application and adoption of the findings in the broader medical community.

ELIGIBILITY:
The study population can be viewed from the cluster (clinic), clinician, staff, or patient level.

At the cluster (clinic) level: To be eligible to participate in this study, a cluster (clinic) must meet all the following criteria:

1. Active participation in the St. Louis Integrated Health Center Network for Community Academic Partnerships.
2. Employment of at least 3 clinicians who commonly manage adult asthma (defined as managing asthma for at least one adult asthma patient, on average, on a weekly basis).
3. Data provided to Azara for data queries, and
4. Willing and able to receive all components of the SMART implementation bundle (i.e., initial educational outreach visit, ongoing practice facilitation/supervision, audit & feedback, and provision of education of patient-level education aides and SMART asthma action plans and monthly operations committee meetings).

At the clinician/clinical staff level:

To be eligible to participate in this study, a clinician/clinical staff member must meet all of the following criteria:

1. Provision of a signed and dated informed consent form.
2. Current state licenses of physician, assistant physician, nurse practitioner, or physician assistant.
3. Regularly cares for adults with asthma (which may include those trained in family medicine, internal medicine, obstetrics/gynecology, and/or specialty medicine).
4. Willing and able to integrate the SMART implementation bundle into their practice.
5. Willing and able to participate for the entire duration of the study, including the pre-implementation, active implementation, and post-implementation periods.
6. Willing to provide data on prescribing patterns and asthma patient outcomes for the duration of the study.

At the patient level:

To be eligible to participate in this study, a patient must meet all of the following criteria:

1. Age ≥12 years old
2. Diagnosis of asthma, of any severity, coded (i.e., International Classification of Diseases [ICD]-10-CM: J45**).
3. The patient has had ≥2 asthma exacerbations in the last year during which systemic corticosteroids were prescribed, and/or the encounter contains an active prescription for an inhaler that is congruent with medium-dose (or higher) maintenance inhaled corticosteroids (ICS) inhalers or low-dose (or higher) ICS-long-acting β-agonist (LABA) inhalers with concomitant reliever short-acting β-agonist inhalers.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2026-01-06 (Actual); Primary Completion 2027-11-15 (Estimated); Study Completion 2028-11-15 (Estimated)

PRIMARY OUTCOMES:
Patient-level Effectiveness (of the SMART implementation bundle) | Through study completion, up to 24 months
  A clinic-level assessment of the SMART implementation bundle with the endpoint of between-group difference in the proportion of SMART-recommended asthma encounters, wherein SMART was the prescribed inhaler regimen. Patient encounters wherein any diagnosis of asthma was coded in patients ≥12 years old will be queried. Asthma encounters will then be in a binary fashion, as either "SMART- non-recommended" or "SMART- recommended" based on asthma exacerbation history and currently prescribed maintenance inhaler medications. A SMART prescription will be defined as clinician prescription of budesonide- formoterol 160/4.5µg or mometasone-formoterol 100/6µg ordered for maintenance and reliever usage. The proportion of SMART prescriptions will be compared between control and intervention groups. The control period will include pre-intervention data, while the intervention period will include all time post-implementation, but exclude the first month as a "transition phase."
Clinician-level adoption (of the SMART implementation bundle) | Through study completion, up to 24 months
  Proportion of clinicians who initially utilize the 3 SMART implementation bundle components. Adoption will be defined by initial: 1) participation in an education and practice facilitation session, 2) participation in an audit and feedback session, 3) use of the patient-centered education aide and action plan, and 4) participation in monthly operations committee meetings. Eligible clinicians will be defined as any clinician that is (1) a currently state-licensed physician, assistant physician, nurse practitioner, or physician assistant, and (2) regularly cares for adults with asthma (defined as managing asthma for at least one adult asthma patient, on average, on a weekly basis).

SECONDARY OUTCOMES:
Clinic-level reach (of the SMART implementation bundle) | Through study completion, up to 24 months
  Number and proportion of eligible clinics that participated in any component of SMART implementation. Clinics will be counted as reached if they participated in any component the SMART implementation bundle. Clinics at partnering clinic systems will be considered potentially eligible for implementation if they cared for ≥100 individuals ≥12 years old with asthma (ICD 10-CM: J45.xx) in the calendar year prior to implementation (2024). Clinic network leadership in coordination with the study steering committee will choose two individual clinic sites within their network they believe to have the highest readiness for SMART implementation.
Clinician-level reach (of the SMART implementation bundle) | Through study completion, up to 24 months
  Number and proportion of eligible clinicians that participated in any component of SMART implementation bundle. Clinicians will be counted as reached if they participated in any component of the SMART implementation bundle (education, practice facilitation, audit and feedback, and/or self-reported use of the asthma action plan or training materials and monthly operations committee meeting at each site) during the active implementation period, which is inclusive of the initial visit and all follow-up visits. A clinician will be considered potentially eligible for SMART implementation (and as such counted as potentially able to be reached) if they are both (1) a physician, nurse practitioner, or physician assistant and (2) have cared for ≥10 adolescents or adults with asthma in the year prior to implementation. This is expected to be inclusive of, but not necessarily limited to, those working in primary care, pediatric, pulmonology, allergy, and/or obstetrics and gynecology clinics.
Staff-level reach (of the SMART implementation bundle) | Through study completion, up to 24 months
  Number and proportion of eligible staff that participated in any component of the SMART implementation bundle. Clinic staff will be counted as reached if they participated in any component of the SMART implementation bundle (education, practice facilitation, audit and feedback, and/or self-reported use of the asthma action plan or training materials and monthly operations committee meeting at each site) during the active implementation period, which is inclusive of the initial visit and all follow-up visits. A clinic staff will be considered potentially eligible for the SMART implementation (and as such counted as potentially able to be reached) if they: (1) provide or may provide clinical advice, and (2) interact with adolescents or adults with asthma, in the opinion of the site CMO and/or site champion. This is expected to be inclusive of, but not necessarily limited to, nursing staff, medical assistants, pharmacists, respiratory therapists, and/or pharmacy techs.
Patient-level reach of (of the evidence-based practice, i.e., SMART) | Through study completion, up to 24 months
  Number of patients with moderate-to-severe asthma prescribed SMART. Patients will be considered to be reached if they were ever prescribed SMART during the active implementation period. A prescription for SMART will count as any script for an ICS-formoterol at the 2024 GINA-recommended dosing on a maintenance and reliever basis. Patients eligible for reach will include any patient age ≥12 years who meets the study- defined definition of moderate-to-severe asthma.
Patient-level effectiveness (of the evidence-based practice, i.e., SMART) | Through study completion, up to 24 months
  Between group difference in the rate of sthma exacerbations. Asthma exacerbations will be defined by: (1) prescription of a new systemic corticosteroid within 7 days of a clinic/telephone encounter for asthma, and/or (2) ICD-10 coding for an acute asthma exacerbation.
Patient-level safety (of the evidence-based practice, i.e., SMART) | Through study completion, up to 24 months
  Between group difference in rate of dysphonia, oral candidiasis, tremor, and/or palpitations and othere reported serious adverse events. Patients will be monitored for serious adverse events and adverse events of special interest (i.e. known side effects of ICS-formoterol by identifying cases of oral candidiasis (thrush; ICD- 10CM: B37.0), dysphonia (ICD-10-CM: R49.0), tremor (ICD-10-CM: R25.1, G25.0, G25.2), or palpitations (R00.2). Clinicians will be asked if they have identified any serious adverse events or adverse events of special interest at site visits during the implementation period. Clinicians will also be provided with the study team's contact information including email and phone number for reporting.
Clinician-level effectiveness (of the SMART implementation bundle) | Through study completion, up to 24 months
  The proportion of clinicians who are "frequent SMART prescribers" (defined as prescribing SMART in ≥30% of indicated encounters). A prescription for SMART will count as script for an ICS- formoterol on a maintenance and reliever basis. Clinicians will be considered eligible if they are both: (1) a physician, nurse practitioner, or physician assistant, and (2) managed ≥10 patients with moderate-to-severe asthma in the year prior to implementation. This is expected to be inclusive of, but not necessarily limited to, those working in primary care, pediatric, pulmonology, allergy, and/or obstetrics and gynecology clinics.
Qualitative assessment (of the SMART implementation bundle and evidence based practice, i.e., SMART) adoption | Through study completion, up to 24 months
  Interviews/focus groups (clinicians, staff) for reasons clinicians/staff participated in implementation components (e.g., time constraints). A subset of clinic leadership, clinicians, and staff will be invited to participate in semi-structured one-on-one interviews (and/or focus groups) regarding reasons for participation and adoption of the implementation bundle.
Clinician-level fidelity to the SMART implementation bundle | Through study completion, up to 24 months
  Proportion of clinicians that participate in both baseline visit and >50% of practice facilitation and audit and feedback sessions.
Clinician-level fidelity (of the evidence-based practice, SMART) | Through study completion, up to 24 months
  Proportion of encounters prescribed SMART intervention as recommended at the correct dose and with SABA inhalers discontinued.
Other system-level implementation outcomes (of the SMART implementation bundle and evidence-based practice, i.e., SMART) | Through study completion, up to 24 months
  Exploratory assessment of costs by the investigators team to implement SMART implementation bundle and cost of asthma management to the payors. A preliminary assessment of estimated cost of training, implementation, asthma morbidity, inhalers and other associated costs will be guided by the Good Practice for Budget Impact Analysis Taskforce recommendations and use cost data from MO HealthNet and the Medical Expenditure Panel Survey.
Patient-level sustainment (of the evidence-based practice, i.e., SMART) | Through study completion, up to 24 months
  Proportion of indicated encounters wherein SMART was prescribed and rate of asthma exacerbations during sustainment vs. intervention period. Maintenance will be assessed by comparing 1) the prescription of SMART and 2) exacerbation rates in the implementation period vs. sustainment period.
Clinician-level and system-level sustainment (of the SMART implementation bundle) | Through study completion, up to 24 months
  A validated sustainability survey will be administered to clinic staff, the site champion, and CMO at each site at the beginning of the sustainment period. At the conclusion of the sustainment period, site champions and CMOs will be given a survey querying how often SMART implementation components were continued during the sustainment period. A

OTHER OUTCOMES:
Qualitative assessment of the determinants of clinician and staff-reach (of the SMART implementation bundle) | Through study completion, up to 24 months
  Reasons clinicians and staff decided to, or decided not to, participate in any component of the SMART implementation bundle. All clinic leadership, clinicians, and staff who were potentially eligible for reach will be invited to complete a survey on why they did (or did not) participate in any component of the SMART implementation bundle. A subset of clinic leadership, clinicians, and staff will be invited to participate in semi- structured one-on-one interviews (and/or focus groups) regarding the reasons they did, or did not, participate in any component of the SMART implementation bundle.
Qualitative assessment of the determinants of clinician and staff-reach (of the evidence-based practice, i.e., SMART | Through study completion, up to 24 months
  Reasons patients decided to or decided not to use SMART. A subset of patients prescribed SMART will be invited to participate in semi- structured one-on-one interviews (and/or focus groups) regarding the reasons they did or did not use SMART.
Reach (of SMART implementation materials including the CHEST website and SMART focused AAP) | Through study completion, up to 24 months
  Number of times CHEST website is visited, and number of times SMART AAP is downloaded from the website. The investigators will describe how often the CHEST website (chestasthmastudy.wustl.edu) is reached by the public and the number of times the SMART AAP is downloaded.
Qualitative assessment (of the SMART implementation bundle and evidence-based practice, i.e., SMART) effectiveness | Through study completion, up to 24 months
  Interviews with clinicians, and staff on effects of the SMART implementation (e.g., workflow, knowledge, self- efficacy) an SMART prescription. All clinic leadership, clinicians, and staff who were potentially eligible for reach will be invited to complete a survey on other effects of the SMART implementation bundle. A subset of clinic leadership, clinicians, and staff will be invited to participate in semi- structured one-on-one interviews (and/or focus groups) regarding other effects of the SMART implementation bundle.
Qualitative assessment (of the SMART implementation bundle and evidence based practice, i.e., SMART) effectiveness | Through study completion, up to 24 months
  Interviews with patients on effects of SMART implementation (i.e., workflow, knowledge, self- efficacy) and SMART prescription. A subset of patients will be invited to participate in semi- structured one-on-one interviews (and/or focus groups) regarding other effects of the SMART implementation bundle.

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - Affinia healthcare, 2220 Lemp Ave, St Louis, Missouri
  - Affinia healthcare, 1717 Biddle Street, St Louis, Missouri
  - Affinia healthcare, 4414 North Florissant Avenue, St Louis, Missouri
  - Family Care Heath Center, 4352 Manchester Ave, St Louis, Missouri
  - Washington University in St. Louis School of Medicine, St Louis, Missouri
  - Family Care Heath Center, 401 Holly Hills Ave, St Louis, Missouri
  - Affinia healthcare, 3396 Pershall Road,, St Louis, Missouri

IPD SHARING:
Plan to Share IPD: Yes
Yes. De-identified IPD will be shared, including quantitative data (demographics, validated surveys, attendance logs, and de-identified EHR data on asthma encounters, diagnoses, and prescriptions) and qualitative interview and focus group transcripts verified for accuracy and de-identified. The protocol, statistical analysis plan, data dictionary, and analytic code will also be shared via NHLBI's BioLINCC. Data will be securely stored within WUSM REDCap, RIS, or Box prior to sharing. HIPAA-compliant transcription and REDCap validation ensure accuracy. Oversight and compliance will be maintained through WUSM IRB, the Office of Information Security, community health center regulatory bodies, and the study's DSMB. Data will follow COREQ, CONSORT, and TIDieR standards and be shared following primary publication.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: De-identified IPD and supporting materials will be submitted to NHLBI's BioLINCC within 12 months after completion of data collection or prior to primary publication, whichever comes first. Data will undergo quality and compliance review before public release. Shared data will remain archived and accessible for long-term preservation within BioLINCC, consistent with NIH and NHLBI repository practices, to enable future secondary analyses and replication studies.
Access Criteria: De-identified IPD and supporting materials will be shared through NHLBI's BioLINCC repository. Access will be open to qualified investigators without restriction for research, replication, or secondary analyses consistent with the study's aims and public health interests. Privacy and confidentiality protections will be maintained per approvals from the WUSM IRB, Office of Information Security, community health center regulatory bodies, and the study's DSMB. Data requests will be reviewed and managed through BioLINCC's standard procedures, which require submission of a data request and execution of a Research Materials Distribution Agreement. Oversight of compliance and continued protection of participant confidentiality will be ensured through WUSM and NHLBI regulatory oversight mechanisms.

REFERENCES:
- [Background] Ivers N, Jamtvedt G, Flottorp S, Young JM, Odgaard-Jensen J, French SD, O'Brien MA, Johansen M, Grimshaw J, Oxman AD. Audit and feedback: effects on professional practice and healthcare outcomes. Cochrane Database Syst Rev. 2012 Jun 13;2012(6):CD000259. doi: 10.1002/14651858.CD000259.pub3. PMID 22696318
- [Background] Infante AF, Wells C, Loza J, Hobbs K, Jarrett JB, Elmes AT. Be SMART About Asthma Management: Single Maintenance and Reliever Therapy. J Am Board Fam Med. 2024 Jul-Aug;37(4):745-752. doi: 10.3122/jabfm.2023.230456R1. PMID 39455262
- [Background] Chapman KR, Barnes NC, Greening AP, Jones PW, Pedersen S. Single maintenance and reliever therapy (SMART) of asthma: a critical appraisal. Thorax. 2010 Aug;65(8):747-52. doi: 10.1136/thx.2009.128504. Epub 2010 Jun 27. PMID 20581409
- [Background] Reddel HK, Bateman ED, Schatz M, Krishnan JA, Cloutier MM. A Practical Guide to Implementing SMART in Asthma Management. J Allergy Clin Immunol Pract. 2022 Jan;10(1S):S31-S38. doi: 10.1016/j.jaip.2021.10.011. Epub 2021 Oct 16. PMID 34666208
- [Background] Norris MR, Modi S, Al-Shaikhly T. SMART - is it practical in the United States? Curr Opin Pulm Med. 2022 May 1;28(3):245-250. doi: 10.1097/MCP.0000000000000862. Epub 2022 Feb 7. PMID 35131990
- [Background] Krings JG, Sekhar TC, Chen V, Blake KV, Sumino K, James AS, Clover AK, Lenze EJ, Brownson RC, Castro M. Beginning to Address an Implementation Gap in Asthma: Clinicians' Views of Prescribing Reliever Budesonide-Formoterol Inhalers and SMART in the United States. J Allergy Clin Immunol Pract. 2023 Sep;11(9):2767-2777. doi: 10.1016/j.jaip.2023.05.023. Epub 2023 May 26. PMID 37245736
- [Background] Zaeh SE, Zimmerman ZE, Eakin MN, Chupp G. Adoption and implementation of maintenance and reliever therapy for adults with moderate-to-severe asthma. Ann Allergy Asthma Immunol. 2024 Sep;133(3):318-324. doi: 10.1016/j.anai.2024.06.011. Epub 2024 Jun 17. PMID 38897404